CLINICAL TRIAL: NCT02616705
Title: Bile Usefulness for Detecting IgG4-related Sclerosing Cholangitis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Nagoya University (Other)
Responsible Party: Principal Investigator, Lewis R. Roberts, Principal Investigator, Mayo Clinic
Other Study IDs: 15-004819
Record Dates: First submitted 2015-11-23; First posted 2015-11-30 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: IgG4-related Sclerosing Cholangitis; IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Bile
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IgG4-related sclerosing cholangitis: Patients with IgG4-related sclerosing cholangitis (also called IgG4 associated cholangitis, IgG4 related cholangitis, or biliary IgG4-related disease)
- Controls: cholangiocarcinoma, PSC, and other patients with biliary strictures

SUMMARY:
Immunoglobulin G4-related disease (IgG4-RD) is an uncommon inflammatory disorder that may affect multiple organ systems, including the biliary tree. IgG4-sclerosing cholangitis (IgG4-SC) can be difficult to distinguish from primary sclerosing cholangitis (PSC) or cholangiocarcinoma (CCA). The investigators aim to evaluate the sensitivity and specificity of bile for the diagnosis of IgG4-SC. Bile samples of patients with biliary strictures of various causes, including IgG4-SC, PSC, and CCA, will be collected during clinical cholangiography procedures. IgG4 will be measured in bile specimens and bile IgG4 concentrations compared between IgG4-SC, PSC, CCA, and other types of biliary strictures.

DETAILED DESCRIPTION:
This study will recruit cases from Mayo Clinic Rochester and Japanese institutions such as Nagoya City University Hospital, Nagoya Daini Red Cross Hospital, and Kurashiki Central hospital. Participants will be individuals who will receive endoscopic retrograde cholangiography (ERC), endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) or percutaneous transhepatic cholangiography (PTC). Bile samples collected from the target cases will be assayed for IgG4 concentration.

ELIGIBILITY:
Inclusion Criteria:

* The presence of a biliary stricture
* 18 years and older
* Consented to IRB 707-03

Exclusion Criteria:

* Younger than 18 years of age
* Unable to collect a bile sample
* Abnormal postsurgical anatomy preventing collection of a bile sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases with biliary stricture(s) of any cause
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2015-11; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Ability of bile IgG4 concentration to distinguish between IgG4-SC, PSC, and CCA. | 2 year
  Bile concentration of IgG4 will be measured in cases and controls, and the groups will be compared using appropriate statistical methods

SECONDARY OUTCOMES:
Correlation between bile and serum IgG4 concentrations. | 2 years
  The relationship between Bile and serum IgG4 concentrations will be assessed for case and controls, using appropriate statistical methods

CONTACTS AND LOCATIONS:
Overall Officials: Lewis R Roberts, MB, ChB, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Nagoya City Universty Graduate School of Medical Sciences, Nagoya, Japan

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing could be arranged and will require IRB approval

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials